CLINICAL TRIAL: NCT05302947
Title: Tocilizumab, Netakimab, and Baricitinib Versus Standard of Care Therapy in Patients With Mild to Moderate COVID-19 - a Retrospective Observational Study
Brief Title: COVID-19 Study at the Russian Clinical and Research Center of Gerontology of the Pirogov RNRMU
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Collaborators: City Clinical Hospital No.52 of Moscow Healthcare Department (Other)
Responsible Party: Principal Investigator, Dmitry Chudakov, Professor Chudakov D.M., D.Sc., Director of Research Institute of Translational Medicine, Head of the Department of molecular technologies, Pirogov Russian National Research Medical University
Other Study IDs: BaToNe-COV-2; 075-15-2020-807 (Other Grant/Funding Number: Ministry of Science and Higher Education RF)
Record Dates: First submitted 2022-03-29; First posted 2022-03-31 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Mild to Moderate
Keywords: tocilizumab; baricitinib; netakimab; anti-IL-17; c-reactive protein; lactic dehydrogenase; neutrophil-to-lymphocyte ratio
MeSH Terms: conditions — COVID-19 | interventions — baricitinib; tocilizumab; netakimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Baricitinib: group included patients received Baricitinib in addition to standard of care therapy
  Interventions: Drug: Baricitinib Oral Tablet
- Tocilizumab: group included patients received Tocilizumab in addition to standard of care therapy
  Interventions: Drug: Tocilizumab Injection
- Netakimab: group included patients received Netakimab in addition to standard of care therapy
  Interventions: Drug: Netakimab
- Control: group included patients received only standard of care therapy at the time of hospital admission according to the corresponding COVID-19 Russian guidelines 2020.
  Interventions: Other: Standard of care therapy

INTERVENTIONS:
Drug: Baricitinib Oral Tablet — Baricitinib was administered at a dose of 4 mg once or twice per day for 3-8 days (5 days on average) depending on the individual patients' condition
  Other Names: Olumiant
  Groups: Baricitinib
Drug: Tocilizumab Injection — Tocilizumab was administered by a single intravenous dose of 400 mg
  Other Names: Actemra
  Groups: Tocilizumab
Drug: Netakimab — Netakimab was administered by a single subcutaneous injection of 120 mg
  Other Names: Efleira
  Groups: Netakimab
Other: Standard of care therapy — SOC treatment included hydroxychloroquine (400 mg twice on day 1, followed by 200 mg twice per day on days 5-10), azithromycin (500 mg once per day for 5 days), lopinavir-ritonavir (400/100 mg twice per day for 14 days), and low molecular-weight heparin according to personal indicators
  Other Names: SOC
  Groups: Control

SUMMARY:
This is a retrospective observational cohort study. About 1000 hospital charts of adult patients admitted to the hospital with mild-to-moderate COVID-19 from February to August 2020 were analyzed to evaluate the inflammatory markers and clinical outcomes.

The aim of this study was to compare the observed results of targeted immunosuppressive therapy, anti-IL-6R (Tocilizumab), anti-IL-17A (Netakimab), and JAK1/JAK2 inhibitor (Baricitinib), with standard-of-care (SOC) therapy. The investigators hypothesize that, as compared to SOC therapy, all target drugs will demonstrate at least similar beneficial effects.

This observation may additionally support a rational choice for mild-to-moderate COVID-19 treatment strategy, considering the general safety profile and patient-specific limitations.

DETAILED DESCRIPTION:
The clinical data from 154 patients were retrospectively collected according to Inclusion and Exclusion criteria. Finally all patients were divided into four groups depending on therapy: 38 patients who received Baricitinib and SOC; 34 patients who received Tocilizumab and SOC; 48 patients who received Netakimab and SOC and 34 patients who received only SOC.

For all patients the investigators assessed the National Early Warning Score2 (NEWS2), absolute neutrophil count (ANC), absolute lymphocyte count (ALC) and blood neutrophil-to-lymphocyte ratio (NLR) at baseline (0 h, the day of therapy started) and after 72 hours (3 days) and 120 hours (5 days) of therapy. The individual dynamics of c-reactive protein (CRP) and lactate dehydrogenase (LDH) were assessed for patients with known parameters at baseline and 72 h (Δ0-72) or at baseline and 120 h (Δ0-120) to avoid excluding from the analysis patients who lacked CRP or LDH data at one of the time points. The individual dynamics of CRP and LDH for patients for whom the results of sequential measurements were available for all three time points was also assessed separately.

Additionally, the clinical outcomes (death or hospital discharge) and amount of days in hospital after starting therapy were estimate for all 154 patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria were included in the study:

1. Patients were hospitalized in two Moscow specialized COVID-19 care units from 02/01/2020 to 08/31/2020.
2. Patients had symptoms of acute respiratory infection (fever, muscle pain, cough) and radiologically-defined viral pneumonia as assessed by computed tomography
3. All patients written informed consent for 'off-label' drug use for persons who received tocilizumab, netakimab, or baricitinib

Exclusion Criteria:

Subjects who meet any of the following criteria were excluded from participation in the study:

1. Pregnant women
2. Patients with unknown National Early Warning Score 2 (NEWS2) metric or with NEWS2 > 6 points on the first day of therapy
3. Patients with the plasma level of CRP > 140 mg/l on the first day of therapy
4. Information about the outcome of patients (death or discharge from the hospital) was absent
5. Patients who first time got the investigational drug later than 72 hours after hospitalization
6. Patients who received a combination of the investigational drugs or application was differed to study design
7. Patients with severe hematological, renal, or liver function impairment or evidence of concomitant bacterial infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed COVID-19, hospitalized into the Russian Clinical and Research Center of Gerontology of the Pirogov RNRMU or the City Clinical Hospital No. 52 of the Department of Health of the City of Moscow from 02/01/2020 to 08/31/2020.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changing in the level of C-reactive protein | 5 days
  The level of C-reactive protein (mg/L ) was measured by ELISA on the day of the start of therapy and then after 72 hours and 120 hours

SECONDARY OUTCOMES:
Changing in the level of Lactate dehydrogenase | 5 days
  The blood level of lactate dehydrogenase (LDH, U/L) was estimate by enzymatic UV-Kinetic method on the day of the start of therapy and then after 72 hours and 120 hours.
Assessment of the absolute lymphocyte count in dynamic | 5 days
  The absolute lymphocyte count (ALC) was assessed by using an automatic hematology analyzer on the day of the start of therapy and then after 72 hours and 120 hours.
Assessment of the absolute neutrophil count in dynamic | 5 days
  The absolute neutrophil count (ANC) was assessed by using an automatic hematology analyzer on the day of the start of therapy and then after 72 hours and 120 hours.
Assessment of the neutrophil-to-lymphocyte ratio | 5 days
  The mathematical ratio of ANC to ALC were calculated for timepoints 0 ( the day of the start of therapy), 3 (72 hours after the start of the therapy) and 5 (120 hours after the start of the therapy)
Changing of the National Early Warning Score2 | 5 days
  The National Early Warning Score2 (NEWS2) metric based on physiological variables including blood pressure, heart rate, respiratory rate, temperature, oxygen saturation, and level of consciousness and falls on a scale of 0 to 20. NEWS2 value at 0-4 points corresponds to low clinical risk, 5-6 points to medium risk and 7 or more points to high clinical risk. NEWS2 was estimate on the day of the start of therapy and then after 72 hours and 120 hours.

OTHER OUTCOMES:
Hospital discharge day and mortality data | 21 days
  The amount of days in the hospital after the start of therapy was estimated for each patients and and analysed as the following groups: less than 4 days in hospital; 5-7 days in hospital; 8-14 days in hospital; more than 15 days in hospital. Outcome (hospital discharge or death) was assessed on the last day of follow-up, the longest period of hospitalisation was 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Zinaida Yu Mutovina, MD-PhD, Principal Investigator — City Clinical Hospital No.52 of Moscow Healthcare Department
Locations (2):
- Russia (2):
  - City Clinical Hospital No. 52 of the Department of Health of the City of Moscow, Moscow
  - Pirogov Russian National Research Medical University, Moscow

IPD SHARING:
Plan to Share IPD: No